CLINICAL TRIAL: NCT00940446
Title: A Comparison of INSORB Staples With Metal Staples in Total Hip Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Orthopaedic Research Foundation (Other)
Collaborators: OrthoIndy (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: DAF_PC000001
Record Dates: First submitted 2009-07-14; First posted 2009-07-16 (Estimated); Results first posted 2018-01-30 (Actual); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Erythema; Drainage; Bruising; Pain
Keywords: Insorb staples; Metal Staples
MeSH Terms: conditions — Erythema; Contusions; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Insorb staples (Experimental): Subcuticular Absorbable staples
  Interventions: Device: Insorb staples
- Control (Active Comparator): Metal staple wound closure
  Interventions: Device: metal staples (Ethicon metal stapler)

INTERVENTIONS:
Device: Insorb staples — absorbable staples required for wound closure
  Other Names: Insorb absorbable stapler; GDW
  Arms: Insorb staples
Device: metal staples (Ethicon metal stapler) — wound closure with metal staples
  Other Names: Ethicon metal stapler
  Arms: Control

SUMMARY:
The purpose of this study is to compare the use of INSORB absorbable staples with metal staples on surgical incision healing after total hip replacement. The study evaluates wound healing, complications, and patient satisfaction regarding wound comfort and appearance after surgery.

DETAILED DESCRIPTION:
Subcuticular closure of wounds can provide superior results to percutaneous suture closure due to the elimination of suture or staple tracts. These tracts can lead to infection and migration of epithelial cells adding to scarring, and cross-hatching scars which remain after healing. Absorbable staples can provide a rapid, secure, subcuticular closure of skin as an alternative to the traditional, manual staple or suture closure. This study will compare INSORB absorbable staples to externally applied standard metal staples with respect to effectiveness of incision closure, acute healing, subject comfort level, security and appearance after total hip replacement.

ELIGIBILITY:
Inclusion Criteria:

* Patient is 18 years or older
* Patient or legal representative is able to understand and provide signed consent for the procedure
* Patient is willing and able to return for required follow-up visits
* Patient needs a total hip arthroplasty surgical procedure

Exclusion Criteria:

* Patient has an active infection
* Patient is enrolled in another similar study
* Patient has a known history of hepatitis
* Patient has a known history of HIV
* Patient has a known history of AIDs
* Patient has a known history of IV drug abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2007-07; Primary Completion 2010-04-30 (Actual); Study Completion 2010-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David A Fisher, MD, Principal Investigator — Indiana Orthopaedic Hospital
Locations (1):
- Indiana Orthopaedic Hospital, Indianapolis, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Insorb Staples: Subcuticular Absorbable staples
  Each participant will have a measured BMI, a measured incision length and documented number of Insorb staples placed. At hospital discharge, 10 days post operatively and 6 weeks postoperatively, each participant will be evaluated for overall wound appearance, intactness of incision, gaping in the incision area, redness at the incision site, swelling at the incision site, a description of the surrounding tissue by the surgeon, documentation of incisional crusting, or fluid exudation. Any palpation or protrusion of the Insorb staple will be documented and patients will be asked to rate comfort and pain related to the Insorb staples.
- Control: Metal staple wound closure
  Each participant will have a measured BMI, a measured incision length and documented number of metal staples placed. At hospital discharge, 10 days post operatively and 6 weeks postoperatively, each participant will be evaluated for overall wound appearance, intactness of incision, gaping in the incision area, redness at the incision site, swelling at the incision site, a description of the surrounding tissue by the surgeon, documentation of incisional crusting, or fluid exudation. Patients will be asked to rate comfort and pain related to the metal staple wound closure.
Period: Overall Study
Arm/Group | Insorb Staples | Control
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Insorb Staples | Control | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Median (Full Range); unit: years] | 62.3 [45 to 82] | 61.9 [41 to 82] | 61.9 [41 to 82]
Sex: Female, Male [Count of Participants; unit: Participants] — number and sex of study participants
  Participants
    Female | 15 | 20 | 35
    Male | 15 | 10 | 25
Number of staples placed [Number; unit: staples] — we counted the number of staples used, collectively for all participants. This is a baseline number used for outcomes comparisons.
  staples | 465 | 597 | 1062

OUTCOME MEASURES:

1. Primary Outcome: Participants With Incisional Drainage, Swelling or Gaps of Incision
Description: Incisional drainage, swelling, gaps of incision. Drainage and swelling will be objectively determined by investigator. Gaps will be measured in millimeters.
Time Frame: Discharge from initial hospital stay (2-5 days post-op)
Measure: Number; unit: participants
Groups:
- Control-metal Staples: Metal staple wound closure
  Each participant will have a measured BMI, a measured incision length and documented number of metal staples placed. At hospital discharge, 10 days post operatively and 6 weeks postoperatively, each participant will be evaluated for overall wound appearance, intactness of incision, gaping in the incision area, redness at the incision site, swelling at the incision site, a description of the surrounding tissue by the surgeon, documentation of incisional crusting, or fluid exudation. Patients will be asked to rate comfort and pain related to the metal staple wound closure.
Arm/Group | Insorb Staples | Control-metal Staples
Number analyzed (Participants) | 30 | 30
participants | 10 | 16

2. Secondary Outcome: Participants With Wound Complications - Hematoma
Description: Assessment of wound for complications, especially hematomas at 6 weeks post surgery. Participants will be scored based on presence of a hematoma or not.
Time Frame: up to 6 weeks post-op
Measure: Number; unit: participants
Groups:
- Insorb Staples: Subcuticular Absorbable staples
  30 enrollees
  Avg age
  Avg BMI
  Sex
  Avg # staples placed
  Avg incision length
- Control: Metal staple wound closure
  30 enrollees
  Avg age
  Avg BMI
  Sex
  Avg # staples placed
  Avg incision length
Arm/Group | Insorb Staples | Control
Number analyzed (Participants) | 30 | 30
participants | 0 | 1

ADVERSE EVENTS:
Arm/Group | Insorb Staples | Control
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No